CLINICAL TRIAL: NCT00772317
Title: A Multicenter Clinical Study of the Sonablate® 450 (Sonablate) for the TreAtment of Locally Recurrent Prostate Cancer With HIFU (STAR Trial)
Brief Title: A Multicenter Clinical Study of the Sonablate®450 for the TreAtment of Locally Recurrent Prostate Cancer With HIFU (STAR Trial)
Acronym: STAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SonaCare Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FSI-003
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Recurrent Prostate Cancer
Keywords: Recurrent; prostate cancer; ebrt; hifu
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIFU (Experimental): High Intensity Focused Ultrasound
  Interventions: Device: High Intensity Focused Ultrasound

INTERVENTIONS:
Device: High Intensity Focused Ultrasound — High Intensity Focused Ultrasound
  Other Names: Sonablate 450; Sonablate

SUMMARY:
For the treatment of locally recurrent prostate cancer following failed external beam radiation therapy (EBRT)

DETAILED DESCRIPTION:
The proposed study is a non-randomized, prospective, single arm study. The safety and effectiveness of the Sonablate treatment in subjects with locally recurrent prostate cancer will be evaluated with regard to freedom from biochemical failure and disease recurrence following HIFU treatment.

Men with histologically confirmed, locally recurrent, organ-confined, non-metastatic prostatic adenocarcinoma two or more years following EBRT, PSA ≥0.5 ng/mL and ≤10 ng/mL, 40 to 85 years of age, and with initial staging of T1c-T2 prior to radiation, who meet the criteria for salvage treatment, will be enrolled.

This pivotal study will cover pre-treatment through the 12-month post-treatment follow-up visit (8 visits).

A 5 year extended follow-up study will be conducted annually for the 2nd-5th years post treatment (4 additional visits).

ELIGIBILITY:
Inclusion Criteria:

* subjects with initial presentation of organ confined recurrent prostate cancer (Stages T1c and T2 only) who have been treated with EBRT (conventional, 3D conformal, or IMRT) or proton therapy, two or more years prior, and currently have biopsy proven local recurrence. Previous radiation therapy must be a documented therapeutic dose of 60 to 81Gy or GyE (gray equivalent) for proton therapy;
* Negative bone scan within 6 months prior to enrollment to rule out possibility of metastases;
* Negative CT scans of the chest, abdomen, and pelvis within 6 months prior to enrollment to rule out possibility of metastases;
* age ≥40 years through ≤85 years of age;
* prostate biopsy with ≥10 core biopsies demonstrating 1 or more cores positive for cancer cells, within 6 months prior to treatment;
* prostate volume ≤ 40 gms(cc) (HIFU subject prostate volume will be initially calculated utilizing TRUS measurements during screening and verified with the use of the Sonablate before initiating the HIFU procedure. Patients with prostate volumes greater than 40 gm(cc) as determined by either measurement will not be enrolled in the study);
* AP diameter of the prostate must be ≤4.0cm;
* serum prostate specific antigen (PSA) ≥0.5 ng/mL and ≤10 ng/mL;
* >90 days post hormone therapy usages, subjects who have or are currently undergoing hormone therapy (GnRH agonist/antagonist) must discontinue hormone therapy and go through a 90 day washout period prior to consideration for study participation, and must remain off hormone therapy throughout the duration of the follow-up period (5 years);
* signed informed consent for the HIFU treatment study through the 12 month follow-up visit (7 visits) and then through the extended follow-up period of 5 years (4 additional visits);
* life expectancy > 12 months.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) criteria of IV or higher;
* intra-prostatic calcifications >1.0 cm (single or continuous grouping) on 2 or more consecutive images along the same plane by either the TRUS or Sonablate 500 measurement will not be enrolled;
* active, uncorrected bleeding disorder as determined by abnormal prothrombin time, partial thromboplastin time, or INR at the time of HIFU (use international lab normal ranges for parameters);
* use of coumadin or any other anticoagulant, unless anticoagulation can be temporarily reversed or stopped;
* active urinary tract infection;
* interest in future fertility;
* body weight which would preclude proper suprapubic catheter functioning, per investigator's discretion
* inability to visualize the prostatic tissue adequately on transrectal ultrasound imaging;
* use of any 5ARI drugs within 3 months prior to enrollment such as Finasteride (Proscar) or Dutasteride (Avodart);
* a debulking transurethral resection of the prostate (TURP) is not acceptable once the screening biopsy for patient selection has been conducted;
* prior treatment for prostate cancer, other than EBRT or hormone therapy;
* history of urethral stent or urethral surgery (urethral dilation, urethroplasty); a Uroflow exam may be conducted at the investigators discretion;
* prior significant rectal surgery (hemorrhoidectomy is acceptable; rectal resection/fissure repair are excluded);
* history of inflammatory bowel disease of the rectum;
* history of any other malignancy treated within the last 5 years, other than squamous or basal cell skin cancer;
* functional bladder problems defined as IPSS > 19;
* current bladder cancer, urethral stricture, or bladder neck contracture; a cystoscopy my be performed at the investigator's discretion to rule out these conditions;
* urinary tract or rectal fistula;
* rectal fibrosis/stenosis; anoscopy or proctoscopy may be performed at the investigator's discretion;
* anomaly of the rectal anatomy or mucus membrane; anoscopy or proctoscopy may be performed at the investigator's discretion;
* prostate seroma/abscess;
* current symptomatic radiation proctitis requiring creams;
* participation in other investigational studies, unless approved in writing by the study sponsor.

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2008-07; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
absence of biochemical failure, defined as achieving a PSA nadir of ≤ 0.5 ng/mL within 12 months of treatment | 12 months post treatment

SECONDARY OUTCOMES:
negative prostate biopsy at the 12 month time point | 12 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mark Carol, MD, Study Director — SonaCare Medical, LLC
Locations (16):
- United States (14):
  - Tower Urology, Los Angeles, California
  - David Geffen School of Medicine at University of California Los Angeles, Los Angeles, California
  - Walter Reed National Military Medical Center (Military Personnel Only), Washington D.C., District of Columbia
  - Specialists in Urology, P.A., Naples, Florida
  - Indiana University, Indianapolis, Indiana
  - Metropolitan Urology, PSC, Jeffersonville, Indiana
  - Tulane University, New Orleans, Louisiana
  - New York University School of Medicine, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland Case Medical Center, Cleveland, Ohio
  - Urologic Consultants of SE PA, LLP, Bala-Cynwyd, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - CAN-AM, Toronto, Ontario